CLINICAL TRIAL: NCT05514262
Title: The Effect on Pain and Satisfaction of Two Different Non-Pharmacological Methods Used During Coronavirus (Covid-19) Vaccination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, Bursa Uludag University, Department of Nursing, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/15-2
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Individual Satisfaction; Pain Management
Keywords: covid-19; covid-19 vaccine; pain control; nonpharmacological method; satisfaction
MeSH Terms: conditions — Agnosia; COVID-19; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The intervention and measurements were carried out by the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- The stress ball group (Experimental): With this group, a yellow stress ball will be used which is 6cm in diameter, of medium hardness and made of high quality silicone, and which returns to its original shape after being squeezed. The researcher will explain to the individuals in the group how they should use the stress ball five minutes before beginning the vaccination and during the procedure. The individuals will be taught to take the stress ball in their right hand, the side on which the vaccination will not be given, and, counting from one to three, to squeeze and release the ball, continuing until the procedure is finished. It will be explained that during the procedure, they should give their attention to the stress ball and focus on squeezing it.
  Interventions: Other: The stress ball
- The Buzzy® group (Experimental): Individuals in this group will use the Buzzy® device. Before the vaccination procedure, the researcher will place the Buzzy® device, which will be at room temperature, on the vaccination site, and it will vibrate in a non-discomforting way for one minute. After this, the Buzzy® device will be removed from the site, and the nurse will perform the vaccination. Because Buzzy® is a device which can be re-used, it will be disinfected after each vaccination procedure, and re-used with other individuals. The Buzzy® device also has ice wings which will not be used in this study, and only the body of the device will be used to provide vibration.
  Interventions: Device: The Buzzy® device
- The control group (No Intervention): Individuals included in the control group will receive no intervention before the vaccination procedure, and the routine Covid-19 vaccination procedure will be used.

INTERVENTIONS:
Other: The stress ball — Covid-19 vaccination procedure with individuals in the stress ball group: With this group, a yellow stress ball will be used which is 6cm in diameter, of medium hardness and made of high quality silicone, and which returns to its original shape after being squeezed. The researcher will explain to the individuals in the group how they should use the stress ball five minutes before beginning the vaccination and during the procedure. The individuals will be taught to take the stress ball in their right hand, the side on which the vaccination will not be given, and, counting from one to three, to squeeze and release the ball, continuing until the procedure is finished. It will be explained that during the procedure, they should give their attention to the stress ball and focus on squeezing it.
  Arms: The stress ball group
Device: The Buzzy® device — Covid-19 vaccination procedure with individuals in the Buzzy® group: Individuals in this group will use the Buzzy® device. Before the vaccination procedure, the researcher will place the Buzzy® device, which will be at room temperature, on the vaccination site, and it will vibrate in a non-discomforting way for one minute. After this, the Buzzy® device will be removed from the site, and the nurse will perform the vaccination. Because Buzzy® is a device which can be re-used, it will be disinfected after each vaccination procedure, and re-used with other individuals. The Buzzy® device also has ice wings which will not be used in this study, and only the body of the device will be used to provide vibration.
  Arms: The Buzzy® group

SUMMARY:
The aim of this study was to determine the effect on pain and satisfaction during the administration of Covid-19 vaccination of two different non-pharmacological methods: squeezing a stress ball and placing Buzzy® on the injection site.

The research was planned with a prospective, randomized controlled and experimental design. Data collection will take place at the Covid-19 Vaccination Clinic of the Health Research and Application Center of Bursa Uludağ University. The research sample will consist of individuals who on the date of the beginning of the data collection stage asked for or approved the Pfizer-BioNTech vaccination for themselves from the Turkish Ministry of Health, and who agreed to participate in the research.

The size of the study sample was statistically determined with the program G*Power 3.1.7. As a result of power analysis, the total minimum sample width was calculated as 120 people, with 40 in each group, accepting type I error level as 5% and in order to achieve an 80% power level. Individuals who meet the research criteria will be assigned to the implementation and control groups by means of a randomization list created by computer according to age and gender.

Research data will be collected face to face, using an Individual Description Form, a Visual Comparison Scale and a Visual Individual Satisfaction Scale.

The following interventions will be performed on the individuals in the intervention group in addition to the standard vaccination procedure:

Covid-19 vaccination procedure with individuals in the stress ball group: With this group, a yellow stress ball will be used which is 6cm in diameter, of medium hardness and made of high quality silicone, and which returns to its original shape after being squeezed. The researcher will explain to the individuals in the group how they should use the stress ball five minutes before beginning the vaccination and during the procedure. The individuals will be taught to take the stress ball in their right hand, the side on which the vaccination will not be given, and, counting from one to three, to squeeze and release the ball, continuing until the procedure is finished. It will be explained that during the procedure, they should give their attention to the stress ball and focus on squeezing it.

Covid-19 vaccination procedure with individuals in the Buzzy® group: Individuals in this group will use the Buzzy® device. Before the vaccination procedure, the researcher will place the Buzzy® device, which will be at room temperature, on the vaccination site, and it will vibrate in a non-discomforting way for one minute. After this, the Buzzy® device will be removed from the site, and the nurse will perform the vaccination. Because Buzzy® is a device which can be re-used, it will be disinfected after each vaccination procedure, and re-used with other individuals. The Buzzy® device also has ice wings which will not be used in this study, and only the body of the device will be used to provide vibration.

Covid-19 vaccination procedure with individuals in the control group: Individuals included in the control group will receive no intervention before the vaccination procedure, and the routine Covid-19 vaccination procedure will be used.

Immediately after the administration of the vaccination, an assistant researcher who is unaware of the injection method used will ask individuals from all groups to assess their pain levels with the Visual Comparison Scale and their satisfaction with the procedure by means of the Visual Individual Satisfaction Scale, and the scores will be recorded on the data collection forms.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect on pain and satisfaction during the administration of Covid-19 vaccination of two different non-pharmacological methods: squeezing a stress ball and placing Buzzy® on the injection site.

The research was planned with a prospective, randomized controlled and experimental design. Data collection will take place at the Covid-19 Vaccination Clinic of the Health Research and Application Center of Bursa Uludağ University. The research sample will consist of individuals who on the date of the beginning of the data collection stage asked for or approved the Pfizer-BioNTech vaccination for themselves from the Turkish Ministry of Health, and who agreed to participate in the research.

The size of the study sample was statistically determined with the program G*Power 3.1.7. As a result of power analysis, the total minimum sample width was calculated as 120 people, with 40 in each group, accepting type I error level as 5% and in order to achieve an 80% power level. Individuals who meet the research criteria will be assigned to the implementation and control groups by means of a randomization list created by computer according to age and gender. That is, the group in which the individuals are placed will be determined by a randomization method according to a randomization list created on a computer.

Research data will be collected face to face, using an Individual Description Form, a Visual Comparison Scale and a Visual Individual Satisfaction Scale.

Individual Description Form: This form will contain questions on the individual's age, gender, education level, height, weight, and previous Covid-19 vaccinations.

Visual Comparison Scale (VCS): The VCS is a 10-cm-long scale used to assess pain intensity felt during a procedure. One end represents no pain, and the other end the most severe pain possible. In this study, a vertical scale will be used.

Visual Individual Satisfaction Scale: The individuals' state of satisfaction during the administration of the vaccination will be assessed with the Visual Individual Satisfaction Scale, which consists of a 10-cm vertical line, at one end of which is written "I am very satisfied" and at the other "I am not at all satisfied".

Close attention will be paid to Covid-19 precautions when collecting research data. After confirming the voluntary participation of the individuals, they will be assigned to the intervention and control groups. After that, their descriptive characteristics will be recorded on a data collection form, and then they will be given information on the use of the Visual Comparison Scale and the Visual Individual Satisfaction Scale.

All of the individuals will receive the vaccination with the use of the 1-ml syringes distributed specifically for the vaccinations according to the specifications of the Turkish Ministry of Health. All vaccinations will be given to the deltoid muscle as one dose (0.3ml). It is planned that all vaccinations will be administered by the same nurse working in the Vaccination Unit, with individuals in an appropriate sitting position, into the deltoid muscle of the left upper arm at an angle of 90° and without aspiration. Determination of the deltoid area where the vaccination will be administered will be achieved in this way: an imaginary horizontal line will be drawn on the outside surface of the arm to which the vaccination is to be administered to the end of the humerus; each end of this imaginary line will join in the axillary alignment to form an inverted triangle, and the area in the middle of the triangle will be used as the injection area. The standard vaccination administration procedure steps will be followed for all individuals in the intervention and control groups.

The following interventions will be performed on the individuals in the intervention group in addition to the standard vaccination procedure:

Covid-19 vaccination procedure with individuals in the stress ball group: With this group, a yellow stress ball will be used which is 6cm in diameter, of medium hardness and made of high quality silicone, and which returns to its original shape after being squeezed. The researcher will explain to the individuals in the group how they should use the stress ball five minutes before beginning the vaccination and during the procedure. The individuals will be taught to take the stress ball in their right hand, the side on which the vaccination will not be given, and, counting from one to three, to squeeze and release the ball, continuing until the procedure is finished. It will be explained that during the procedure, they should give their attention to the stress ball and focus on squeezing it.

Covid-19 vaccination procedure with individuals in the Buzzy® group: Individuals in this group will use the Buzzy® device. Before the vaccination procedure, the researcher will place the Buzzy® device, which will be at room temperature, on the vaccination site, and it will vibrate in a non-discomforting way for one minute. After this, the Buzzy® device will be removed from the site, and the nurse will perform the vaccination. Because Buzzy® is a device which can be re-used, it will be disinfected after each vaccination procedure, and re-used with other individuals. The Buzzy® device also has ice wings which will not be used in this study, and only the body of the device will be used to provide vibration.

Covid-19 vaccination procedure with individuals in the control group: Individuals included in the control group will receive no intervention before the vaccination procedure, and the routine Covid-19 vaccination procedure will be used.

Immediately after the administration of the vaccination, an assistant researcher who is unaware of the injection method used will ask individuals from all groups to assess their pain levels with the Visual Comparison Scale and their satisfaction with the procedure by means of the Visual Individual Satisfaction Scale, and the scores will be recorded on the data collection forms.

ELIGIBILITY:
Inclusion Criteria:

* Approving the Pfizer-BioNTech vaccination from the Turkish Ministry of Health
* Not having had an injection or vaccination in the deltoid muscle for at least three months
* Participating voluntarily in the study
* Being able to speak and understand Turkish
* Being aged 18 years or older
* Not having any vision or auditory problems
* Not having any condition which might affect pain sensation
* Not having developed any complication which would hinder a delta muscle injection.

Exclusion Criteria:

* Not wanting to participate in the study, or during the course of the research, wishing to withdraw from the study
* Having any condition which would affect the sensation of pain
* Not being able to agree on a place or time
* Being less than 18 years of age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure-1 | 4 months
  pain intensity in mm
Primary Outcome Measure-2 | 4 months
  the individuals' state of satisfaction in mm

SECONDARY OUTCOMES:
Secondary Outcome Measure-1 | 4 months
  weight in kilograms
Secondary Outcome Measure-2 | 4 months
  height in meters
Secondary Outcome Measure-3 | 4 months
  BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Elmas Baki, MSc, Study Chair — Bursa Uludağ University Health Applications Research Center

IPD SHARING:
Plan to Share IPD: No